CLINICAL TRIAL: NCT04130243
Title: Biomarkers in Congenital Heart Diseases and Pulmonary Arterial Hypertension
Brief Title: Biomarkers in Pediatric Congenital Heart Disease and PAH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. R.M.F. Berger, Head of Pediatric Cardiology, University Medical Center Groningen
Other Study IDs: 201700243
Record Dates: First submitted 2017-05-01; First posted 2019-10-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Congenital Heart Disease; Pulmonary Arterial Hypertension
Keywords: Biomarker; Congenital Heart Disease; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Arterial Hypertension | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenital Heart disease: In patients with (a history of) pressure- and/or volume loaded right ventricle due to congenital heart disease extra blood will be withdrawn for a blood test; serumbiomarker
  Interventions: Other: Blood test
- Pulmonary Arterial Hypertension: In patients with (a history of) pressure- and/or volume loaded right ventricle due to pulmonary arterial hypertension extra blood will be withdrawn for a blood test; serumbiomarker
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Withdrawal of (extra) blood to measure serum biomarkers with a blood test

SUMMARY:
Nowadays, biomarkers are broadly used in clinical practice. Blood-derived biomarkers fulfil an important role in the field of cardiology. However, most biomarkers have been investigated for adult left ventricular disease. In congenital heart diseases (CHD) and pulmonary arterial hypertension (PAH), which involves children and mostly the right ventricle, less is known about the clinical and predictive value of blood-derived biomarkers. Since the group of survivors of CHD and PAH is growing because of the improved techniques nowadays, development of better tools to maintain the quality of life for the longer term in these patients is urgently needed. Blood-derived biomarkers are minimally invasive biomarkers, are quantitative and have shown to be able to reveal pathological processes in an early stage. Hence, blood-derived biomarkers may be a good addition to current diagnostic means in CHD and PAH.

Objective: The primary objective of this study is to investigate cross-sectionally the association between various emerging blood-derived biomarkers and right ventricular (RV) function:defined as tricuspid annular plane systolic excursion (TAPSE) measured with echocardiography, in children with (a history of ) an abnormally loaded, volume and/or pressure loaded, right ventricle associated with CHD and/or PAH.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

The primary objective is to investigate cross-sectionally (at baseline and after one year) the association between various emerging blood-derived biomarkers and right ventricular (RV) function:defined as tricuspid annular plane systolic excursion (TAPSE) measured with echocardiography, in children with (a history of ) an abnormally loaded, volume and/or pressure loaded, right ventricle associated with CHD and/or PAH.

TIME FRAME: Baseline and after one year.

Secondary Objective:

Furthermore, the investigators aim to explore:

* The stability, dynamic (treatment-induced) longitudinal changes of these biomarkers and their association with RV function (defined as TAPSE).
* The predictive value of these biomarkers measured at baseline with regard to various clinically relevant impaired RV functioning parameters (TAPSE, RV- Fractional area change , RV-Fractional shortening and RV function assessed with eyeballing) at long term follow-up.
* The predictive value of these biomarkers with regard to clinical outcome defined as the composite of mortality, hospitalization, and or heart/lung transplantation.

STUDY POPULATION: All patients with (a history of) an abnormally loaded right ventricle associated with CHD and/or PAH who are followed in the Center of Congenital Heart Disease - University Medical Center Groningen (CHH-UMCG) from 01-12-2017 will be approached by letter and telephone to be included.

STUDY PROCEDURES:

1. The study is introduced to the patient and his/her parents/legal representatives by letter and telephone. When the patient or his/her parents/legal representatives are interested the researcher will ask them to sign informed consent papers. When the patient is admitted to the clinical ward or will come for his/her outpatient clinic visit the researcher will check if informed consent has been given. If informed consent has been given and the patient meets the inclusion criteria he/she will be included in the study.
2. Study procedures with respect to primary comparison:

   Echocardiography will be performed in all included patients (100%) in context of standard care. Blood drawing in context of standard care or additional study purposes will be performed in all included patients (100%).
3. Study procedures (all performed in context of standard care) with respect to secondary comparisons: Mortality will be assessed in all patients (±100%).Functional class will be clearly documented in most included patients (±80%).MRI will be performed in a subpopulation of included patients (±50%).CPET will be performed in a subpopulation of included patients (±40%). 6MWD will be performed in a subpopulation included patients (±30%).

WITHDRAWAL OF INDIVIDUAL SUBJECTS: Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

REPLACEMENT OF INDIVIDUAL SUBJECTS AFTER WITHDRAWAL: Withdrawal before the first time point will result in exclusion. Withdrawal after the first time point will result in a smaller sample size regarding to follow up, but the data will still be used for the available time points.

PREMATURE TERMINATION: premature termination has no influence on the patients.

ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION:

1. In this study the data will be coded according to a protected key on the general Beatrix Children's Hospital (BKK)-disk. Data will be collected in RedCap or Utopia, which both meet the security requirements according to legislation described by BROK and UMCG.

   All included patients will get a study identification number: BioCHD001, BioCHD002, etc. The order will be in the order of the obtained informed consent. The key will be available at the general BKK-disk for above mentioned investigators and contains the original patient number (UMCG-number), study identification number (study ID), and study identification number of other studies the patient is involved in.

   Data entry will be based on information from Epic, Poliplus, ECHOPAC (for echocardiography) or Medis QMass (for MRI). The blood samples will be stored on study ID by the central laboratory and assessments of the blood-derived biomarkers will be performed by the central laboratory as well. Blood results will be communicated according to study ID.

   Data will be stored in the central laboratory until all the different assays have been run. Data will be kept 15 years after end-of-study. Conditions for long-term document storage will follow GCP, institutional and national guidelines.
2. Monitoring and Quality Assurance : Monitoring will take place according to guidelines in Research Toolbox on UMCG-intranet.
3. Annual progress report: The sponsor/investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.
4. Public disclosure and publication policy: This prospective study will be registered prospectively at the website www.toetsingonline.nl and clintrail.gov.

The results of the study will be published without reservations at international conferences and will be submitted for publication in international "peer-reviewed" scientific journals.

SAFETY REPORTING:

1. Temporary halt for reasons of subject safety:

   In accordance to section 10, subsection 4, of the WMO, the sponsor will suspend the study if there is sufficient ground that continuation of the study will jeopardise subject health or safety. The sponsor will notify the accredited METC without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.
2. Adverse events (AEs) Reporting or recording of adverse events is not applicable in this observational follow up study.
3. The current study is a observational, non-intervention, follow up study in a population that contains patients with possible SAEs as result of their (congenital) heart disease. Therefore, only SAE's resulting from extra blood withdrawals will be reported by the investigator to the sponsor without undue delay after obtaining knowledge of the events.

The sponsor will report the SAEs that are a result of extra blood withdrawal through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 7 days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs, related to extra blood withdrawal, will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

SAMPLE SIZE CALCULATION: In this study the investigators would like to identify blood-derived biomarkers for right ventricular disease in CHD and PAH. In this sample size calculation the investigators have to take into account all the known references of the to be tested biomarkers and that the levels of the biomarkers could differ with respect to age and gender. Previous research confirmed lower levels of specific biomarkers in children compared to adults. Published results concerns mostly significant results with respect to clinically ill versus clinically adapted patients. The investigators would like to look at the correlation between the level of blood-derived biomarkers and RV function. Based on the published results with respect to biomarkers in CHD, a correlation coefficient of (-)0.3 should be sufficient. TAPSE, gender and age are included as predictor variables. With a good prediction level this will give a sample size of 380.

STATISTICAL ANALYSIS PLAN: For the cross-sectionally primary endpoint, the investigators will analyze the correlations of the level of serum biomarker withRV-function (defined as the echocardiographic measurement TAPSE), using Spearman partial correlation analyses, crude and adjusted for age and sex. Subsequently, linear regression analysis will be used to further explore the relationship between biomarkers with continuous RV function. This will be done at baseline and after one year.

For the exploratory objectives, the stability of biomarkers in time will be assessed using intraclass correlation coefficients.Repeated measures linear mixed model techniques will be applied to explore changes of biomarkers and right ventricular function in time in which patients will be entered as the random component of the mixed model. Binary or multinominal logistic regression analysis will be used to assess the relationship between biomarkers and RV function impairment.

Kaplan Meier and Cox regression analysis will be performed to compare (transplantation-free) survival of patients with high or low baseline biomarkers and to explore the predictive value of biomarkers on clinical outcome.

Not normally distributed continous variables (e.g. biomarkers with skewed distribution) will be, if appropriate, log-transformed, prior to inclusion in the regression models.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years
* Patients with Pulmonary Arterial hypertension: diagnosis confirmed according to the standards of the National Expertise Center for PH in childhood.
* Patients with CHD with an abnormally loaded right ventricle including tetralogy of Fallot (TOF), pulmonary (valve) stenosis (PS), pulmonary insufficiency (PI), atrial septal defect (ASD), ventricular septal defect (VSD) and total anomalous pulmonary venous return (TAPVR): diagnosis confirmed by echocardiography or cardiac MRI in UMCG-CCH.

Exclusion Criteria:

* Age >18 years
* Not familiar with Dutch language
* Pregnant
* Concomitant musculoskeletal disease
* No echocardiography available within three months before or after blood collection
* Being under examination for non-diagnosed disease at time of investigation

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population concerns all patients aged 0-18 years with (a history of) an abnormally loaded right ventricle (due to right-sided congenital heart disease or pulmonary arterial hypertension) who visit the outpatient clinic or will be electively admitted at the Center of Congenital Heart Disease - University Medical Center Groningen (CHH-UMCG).
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
TAPSE (mm) TAPSE (tricuspid annular plane systolic excursion) | At baseline (t=0)
  Right ventricular function defined as TAPSE assessed by echocardiography

SECONDARY OUTCOMES:
WHO functional class | At baseline (t=0)
  Disease severity defined as WHO-functional class
WHO functional class | At 1 year
  Disease severity defined as WHO-functional class
Six-minute walk distance (6MWD) | At baseline (t=0)
  Disease severity defined as distance walked at 6MWD
Six-minute walk distance (6MWD) | At 1 year
  Disease severity defined as distance walked at 6MWD
RV fractional area change (RV-FAC) | At 1 year
  Disease severity defined as RV-FAC
RV fractional shortening (RV-FS) | At baseline (t=0)
  Disease severity defined as RV-FS
RV fractional shortening (RV-FS) | At 1 year
  Disease severity defined as RV-FS
RV-function assessed with eyeballing (good, moderate, bad) | At baseline (t=0)
  Disease severity defined RV-function assessed with eyeballing
RV-function assessed with eyeballing (good, moderate, bad) | At 1 year
  Disease severity defined RV-function assessed with eyeballing
NYHA classification | At baseline (t=0)
  Disease severity defined NYHA classification
NYHA classification | At 1 year
  Disease severity defined NYHA classification

OTHER OUTCOMES:
Heart/Lung transplantation per participant | During follow-up of the study; from enrollment till end of the study (5 years later)
  Disease severity defined as undergoing a heart/lung transplantation
Number of Hospitalizations per participant | During follow-up of the study; from enrollment till end of the study (5 years later)
  Hospitalization due to any cause during follow up study
Number of participants that do not survive during follow-up study | During follow-up of the study; from enrollment till end of the study (5 years later)
  Mortality defined as dead due to any cause during follow up study: from enrollment till end of study (5 years later)

CONTACTS AND LOCATIONS:
Overall Officials: A AE Verhagen, MD PhD, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braunwald E. Biomarkers in heart failure. N Engl J Med. 2008 May 15;358(20):2148-59. doi: 10.1056/NEJMra0800239. No abstract available. PMID 18480207
- [Background] Nagarajan V, Hernandez AV, Tang WH. Prognostic value of cardiac troponin in chronic stable heart failure: a systematic review. Heart. 2012 Dec;98(24):1778-86. doi: 10.1136/heartjnl-2012-301779. Epub 2012 Oct 31. PMID 23118345
- [Background] de Boer RA, Daniels LB, Maisel AS, Januzzi JL Jr. State of the Art: Newer biomarkers in heart failure. Eur J Heart Fail. 2015 Jun;17(6):559-69. doi: 10.1002/ejhf.273. Epub 2015 Apr 16. PMID 25880523
- [Background] Kato TS, Armstrong HF, Schulze PC, Lippel M, Amano A, Farr M, Bacchetta M, Bartels MN, Di Tullio MR, Homma S, Mancini D. Left and Right Ventricular Functional Dynamics Determined by Echocardiograms Before and After Lung Transplantation. Am J Cardiol. 2015 Aug 15;116(4):652-9. doi: 10.1016/j.amjcard.2015.05.027. Epub 2015 May 21. PMID 26089014
- [Background] Beghetti M, Berger RM, Schulze-Neick I, Day RW, Pulido T, Feinstein J, Barst RJ, Humpl T; TOPP Registry Investigators. Diagnostic evaluation of paediatric pulmonary hypertension in current clinical practice. Eur Respir J. 2013 Sep;42(3):689-700. doi: 10.1183/09031936.00140112. Epub 2013 Apr 5. PMID 23563261
- [Background] Koch A, Zink S, Singer H. B-type natriuretic peptide in paediatric patients with congenital heart disease. Eur Heart J. 2006 Apr;27(7):861-6. doi: 10.1093/eurheartj/ehi773. Epub 2006 Feb 8. PMID 16467354
- [Background] Van Albada ME, Loot FG, Fokkema R, Roofthooft MT, Berger RM. Biological serum markers in the management of pediatric pulmonary arterial hypertension. Pediatr Res. 2008 Mar;63(3):321-7. doi: 10.1203/PDR.0b013e318163a2e7. PMID 18287971
- [Background] van Loon RL, Roofthooft MT, Delhaas T, van Osch-Gevers M, ten Harkel AD, Strengers JL, Backx A, Hillege HL, Berger RM. Outcome of pediatric patients with pulmonary arterial hypertension in the era of new medical therapies. Am J Cardiol. 2010 Jul 1;106(1):117-24. doi: 10.1016/j.amjcard.2010.02.023. PMID 20609658
- [Background] Takatsuki S, Wagner BD, Ivy DD. B-type natriuretic peptide and amino-terminal pro-B-type natriuretic peptide in pediatric patients with pulmonary arterial hypertension. Congenit Heart Dis. 2012 May-Jun;7(3):259-67. doi: 10.1111/j.1747-0803.2011.00620.x. Epub 2012 Feb 10. PMID 22325151
- [Background] Ploegstra MJ, Douwes JM, Roofthooft MT, Zijlstra WM, Hillege HL, Berger RM. Identification of treatment goals in paediatric pulmonary arterial hypertension. Eur Respir J. 2014 Dec;44(6):1616-26. doi: 10.1183/09031936.00030414. Epub 2014 Jul 17. PMID 25034572
- [Background] Fernandes BA, Maher KO, Deshpande SR. Cardiac biomarkers in pediatric heart disease: A state of art review. World J Cardiol. 2016 Dec 26;8(12):719-727. doi: 10.4330/wjc.v8.i12.719. PMID 28070239
- [Background] Torbicki A, Kurzyna M, Kuca P, Fijalkowska A, Sikora J, Florczyk M, Pruszczyk P, Burakowski J, Wawrzynska L. Detectable serum cardiac troponin T as a marker of poor prognosis among patients with chronic precapillary pulmonary hypertension. Circulation. 2003 Aug 19;108(7):844-8. doi: 10.1161/01.CIR.0000084544.54513.E2. Epub 2003 Aug 4. PMID 12900346
- [Background] Baum H, Hinze A, Bartels P, Neumeier D. Reference values for cardiac troponins T and I in healthy neonates. Clin Biochem. 2004 Dec;37(12):1079-82. doi: 10.1016/j.clinbiochem.2004.08.003. PMID 15589813
- [Background] Reddy S, Bernstein D. Molecular Mechanisms of Right Ventricular Failure. Circulation. 2015 Nov 3;132(18):1734-42. doi: 10.1161/CIRCULATIONAHA.114.012975. PMID 26527692
- [Background] Borgdorff MA, Koop AM, Bloks VW, Dickinson MG, Steendijk P, Sillje HH, van Wiechen MP, Berger RM, Bartelds B. Clinical symptoms of right ventricular failure in experimental chronic pressure load are associated with progressive diastolic dysfunction. J Mol Cell Cardiol. 2015 Feb;79:244-53. doi: 10.1016/j.yjmcc.2014.11.024. Epub 2014 Dec 5. PMID 25486580
- [Background] Pintalhao M, Castro-Chaves P, Vasques-Novoa F, Goncalves F, Mendonca L, Fontes-Carvalho R, Lourenco P, Almeida P, Leite-Moreira A, Bettencourt P. Relaxin serum levels in acute heart failure are associated with pulmonary hypertension and right heart overload. Eur J Heart Fail. 2017 Feb;19(2):218-225. doi: 10.1002/ejhf.611. Epub 2016 Aug 4. PMID 27488261
- [Background] Zelniker T, Uhlmann L, Spaich S, Friedrich J, Preusch MR, Meyer FJ, Katus HA, Giannitsis E. Novel biomarkers for risk stratification in pulmonary arterial hypertension. ERJ Open Res. 2015 Oct 19;1(2):00008-2015. doi: 10.1183/23120541.00008-2015. eCollection 2015 Oct. PMID 27730146
- [Background] Calvier L, Legchenko E, Grimm L, Sallmon H, Hatch A, Plouffe BD, Schroeder C, Bauersachs J, Murthy SK, Hansmann G. Galectin-3 and aldosterone as potential tandem biomarkers in pulmonary arterial hypertension. Heart. 2016 Mar;102(5):390-6. doi: 10.1136/heartjnl-2015-308365. PMID 26869635
- [Background] Knofczynski GT, Mundfrom D. Sample sizes when using multiple linear regression for prediction. Educational and Psychological Measurement. 2008 June; 68(3):431-442.
- [Background] Leberkuhne LJ, Ploegstra MJ, Douwes JM, Bartelds B, Roofthooft MT, Hillege HL, Berger RM. Serially Measured Uric Acid Levels Predict Disease Severity and Outcome in Pediatric Pulmonary Arterial Hypertension. Am J Respir Crit Care Med. 2017 Feb 1;195(3):401-404. doi: 10.1164/rccm.201606-1152LE. No abstract available. PMID 28145758
- [Background] Hartupee J, Mann DL. Positioning of inflammatory biomarkers in the heart failure landscape. J Cardiovasc Transl Res. 2013 Aug;6(4):485-92. doi: 10.1007/s12265-013-9467-y. Epub 2013 May 11. PMID 23666808
- [Background] Webb GD. Challenges in the care of adult patients with congenital heart defects. Heart. 2003 Apr;89(4):465-9. doi: 10.1136/heart.89.4.465. No abstract available. PMID 12639885
- [Background] Norozi K, Zoege M, Buchhorn R, Wessel A, Geyer S. The influence of congenital heart disease on psychological conditions in adolescents and adults after corrective surgery. Congenit Heart Dis. 2006 Nov;1(6):282-8. doi: 10.1111/j.1747-0803.2006.00048.x. PMID 18377495
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Background] Pang PS, Xue Y, Defilippi C, Silver M, Januzzi J, Maisel A. The role of natriuretic peptides: from the emergency department throughout hospitalization. Congest Heart Fail. 2012 Sep-Oct;18 Suppl 1:S5-8. doi: 10.1111/j.1751-7133.2012.00307.x. PMID 22891802